CLINICAL TRIAL: NCT01721902
Title: Stem Cell Implantation in Patients Undergoing CABG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminiated due the lack of recruitment.
Sponsor: Miltenyi Biotec, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0801-133; 808756 (Other: University of Pennsylvania)
Record Dates: First submitted 2012-10-01; First posted 2012-11-06 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Ischemic Cardiomyopathy; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous CD133+ Bone Marrow Stem Cells (Active Comparator): Intra-myocardial injection of autologous CD133+ cells in suspension.
  Interventions: Device: Autologous CD133+ Bone Marrow Stem Cells
- Carrier Solution (Placebo Comparator): Intra-myocardial inception of carrier solution.
  Interventions: Other: Carrier Solution

INTERVENTIONS:
Device: Autologous CD133+ Bone Marrow Stem Cells — Intra-myocardial injection of 2-3 x 10E6 CD133+ Bone Marrow Stem Cells
  Arms: Autologous CD133+ Bone Marrow Stem Cells
Other: Carrier Solution — Intra-myocardial injection of carrier solution
  Arms: Carrier Solution

SUMMARY:
The primary objective of this study is to demonstrate the feasibility and safety of intra-operative, intra-myocardial injection of autologous CD133 positive bone marrow cells at the time of coronary artery bypass graft (CABG) surgery in patients with chronic ischemic cardiomyopathy. Additionally, the feasibility of producing autologous CD133+ bone marrow stem cells will be assessed.

The investigators hypothesize that collection of a sufficient number of CD133+ cells through bone marrow aspiration prior to surgery, with subsequent processing and intra-myocardial injection of high purity cells following completion of CABG, will be feasible without significant adverse clinical consequences.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is the leading cause of death in the U.S. in both men and women and the aging of the population and rising prevalence of diabetes ensure that the number of persons with CHD will continue to increase over the next several decades. Two major factors contributing to adverse outcomes in patients undergoing coronary artery bypass grafting (CABG) surgery are failure to achieve complete revascularization, and residual impairment in left ventricular function.

In the present study, the investigators propose a Phase I randomized double-blind study designed to assess the feasibility and safety of autologous CD133+ cells in patients referred for CABG who have significant regions of viable but non-revascularizable myocardium and/or significant LV systolic dysfunction not likely to improve with conventional coronary revascularization.

Autologous CD133+ bone marrow progenitor cells will be harvested from study subjects at the time of CABG, processed and then injected into patients' myocardium prior to completion of CABG surgery. The test material consists of autologous CD133+ cells. Since intra-myocardial injections per se could stimulate neovascularization, control group patients will receive a placebo injection of carrier solution. Control subjects will thus have an identical procedure to those randomized to autologous CD133+ cell injections.

The three goals of the study are as follows:

1. To demonstrate the feasibility and safety of intra-operative, intra-myocardial injection of autologous CD133+ bone marrow cells in adults with chronic ischemic cardiomyopathy associated with impair left ventricular function.
2. To assess the effect of autologous CD133+ cell injections on regional myocardial perfusion and function by comparing paired magnet resonance scans obtained prior to CABG and again 6 months post CABG.
3. To assess the effect of autologous CD133+ stem cell injections on symptom severity and quality of life at 6 months after CABG surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients with ischemic heart disease manifested by Canadian class II or greater angina and/or New York Heart Association class II, III or IV exercise intolerance AND who have undergone diagnostic coronary angiography demonstrating at least 70% diameter narrowing of at least 2 major coronary arteries or branches or at least 50% diameter narrowing of the left main coronary artery.
* Left ventricular systolic dysfunction evaluated by echocardiography or LV angiography (LV ejection fraction less than or equal to 49%).
* No contraindications or exclusions (see below)
* Willingness to participate and ability to provide informed consent

Exclusion Criteria:

* Contraindications to magnetic resonance imaging .
* Need for emergent revascularization.
* Need for concomitant surgical procedure at the time of CABG (e.g. valve repair or replacement, aneurysm resection, etc.).
* Hemodynamically unstable patients.
* Patients with confirmed transmural myocardial infarction within 4 weeks, and/or rising cardiac biomarker proteins (i.e. troponin), and/or worsening ECG changes.
* Prior CABG surgery.
* Stroke within 1 month prior to planned CABG.
* Diagnosed with human immunodeficiency virus (HIV) or any other immune disorder or immunosuppressive medication (e.g. prednisone, cyclophosphamide, etanercept, etc.)
* Organ dysfunction
* Contra-indication for bone marrow aspiration (Thrombocytopenia < 50.000 mm3, INR > 2.0, use of antiplatelet agents other than aspirin).
* Hemoglobin less than 8g/dL, white blood cell count less than 4,000/mm3, absolute neutrophil count less than 1500/mm3
* Active infection
* Myelodysplastic syndrome (MDS)
* Significant cognitive impairment
* Any condition associated with a life expectancy of less than 6 months
* Patients known allergic reaction or contraindication to any of the component of the CD133+ enriched cells
* Participation in other studies concomitant with this study
* History of severe ventricular tachy-arrythmias
* Inability or unwillingness to provide written informed consent
* Positive serum pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Freedom from a Major Adverse Cardiac Event (MACE) | Six months
  Defined as cardiac death, myocardial infarction (CK/CK-MB over 5 times the upper limit of normal), repeat coronary bypass grafting, or a repeat percutaneous intervention of bypassed coronary artery.
Feedom from any major arrhythmias | Six months
  Defined as sustained ventricular tachycardia or survived sudden death.

SECONDARY OUTCOMES:
Regional myocardial perfusion and function assessed by comparing paired magnetic resonance scans, ECHOs and SPECT scans obtained prior to CABG and again at 6 months post CABG. | 6 months
Symptom severity and quality of life at 6 months after CABG surgery. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ping J Woo, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States